CLINICAL TRIAL: NCT02874846
Title: A Double-masked, Randomized, Placebo-controlled Study of the Nocturnal and Diurnal IOP-lowering Effect of Netarsudil Ophthalmic Solution 0.02% in Habitual Positions Over a 24-hour Period.
Brief Title: Nocturnal/Diurnal Intraocular Pressure-Lowering Effect of Netarsudil Ophthalmic Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS204
Record Dates: First submitted 2016-08-15; First posted 2016-08-22 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2016-10

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — netarsudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Netarsudil Ophthalmic Solution 0.02% (Experimental): 1 drop in each eye (OU) daily
  Interventions: Drug: Netarsudil ophthalmic solution 0.02%
- Netarsudil Ophthalmic Solution Vehicle (Placebo Comparator): 1 drop in each eye (OU) daily
  Interventions: Other: Netarsudil Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: Netarsudil ophthalmic solution 0.02% — Once daily in both eyes (OU) in the evening (PM) for 7 days
  Other Names: AR-13324
  Arms: Netarsudil Ophthalmic Solution 0.02%
Other: Netarsudil Ophthalmic Solution Vehicle — Once daily in both eyes (OU) in the evening (PM) for 7 days
  Arms: Netarsudil Ophthalmic Solution Vehicle

SUMMARY:
To evaluate effect of Netarsudil Ophthalmic Solution 0.02% on Nocturnal and Diurnal Intraocular Pressure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Ocular hypertension or open-angle glaucoma in both eyes.
3. Unmedicated intraocular pressure > 17 mmHg in one or both eyes and < 30 mmHg in both eyes.
4. Corrected visual acuity in each eye equivalent to 20/200 or better.
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

1. Glaucoma with pseudoexfoliation or pigment dispersion component, history of angle closure, narrow angles.
2. Intraocular pressure ≥ 30 mmHg.
3. Use of ocular medications within 30 days.
4. Known hypersensitivity to any component of the test formulations or to medications used routinely during a clinical eye examination.
5. Previous eye surgery (other than cataract).
6. Ocular trauma within 6 months.
7. Clinically significant ocular disease that might interfere with the study.
8. Central corneal thickness greater than 620 µm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals
Locations (1):
- Nancy Ramirez, Bedminster, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peace JH, McKee HJ, Kopczynski CC. A Randomized, Phase 2 Study of 24-h Efficacy and Tolerability of Netarsudil in Ocular Hypertension and Open-Angle Glaucoma. Ophthalmol Ther. 2021 Mar;10(1):89-100. doi: 10.1007/s40123-020-00322-1. Epub 2020 Nov 26. PMID 33244711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who agreed to participate in this study were assessed during a screening visit and those who were already using ocular hypotensive medication had to undergo a washout for a specified period (5 days to 4 weeks, depending on the medication) prior to the Qualification visit.
Groups:
- Netarsudil Ophthalmic Solution 0.02%; Netarsudil Ophthalmic Solution Vehicle: 1 drop in each eye (OU) daily in the evening (PM)
Period: Overall Study
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution Vehicle
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Netarsudil Ophthalmic Solution 0.02%: 1 drop in each eye daily (OU) in the evening (PM)
- Netarsudil Ophthalmic Solution Vehicle: 1 drop in each eye daily (OU) in the evening
- Total: Total of all reporting groups
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.23) | 64.5 (5.07) | 64.4 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) Over Nocturnal Time Period
Description: The primary efficacy endpoint was the mean change from baseline in mean nocturnal IOP (defined as the mean of the 4 nocturnal time points: 21:00, 00:00, 03:00, and 06:00 hours) on Day 8/Day 9
Time Frame: Assessed over 24 hours at 9 pm, midnight, 3 am and 6 am on days 1/2 and 8/9
Population: ITT
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Netarsudil Ophthalmic Solution Vehicle: 1 drop in each eye (OU) daily in the evening
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution Vehicle
Number analyzed (Participants) | 8 | 4
mmHg
  Baseline (Day 1/2); nocturnal mean | 22.84 (2.21) | 23.56 (1.94)
  Visit 4 (Day 8/9); nocturnal mean | 19.38 (2.86) | 23.19 (1.95)

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: 7 days (day 1/2 to day 8/9)
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution Vehicle
Number analyzed (Participants) | 8 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 7 days from day 1/2 to day 8/9.
Arm/Group | Netarsudil Ophthalmic Solution 0.02% | Netarsudil Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No